CLINICAL TRIAL: NCT05876468
Title: " Effects of Continuous Anterior Chest Compression (CACC) & Comparision With Prone Position in ARDS Patients " The StrapVent Study "
Brief Title: Effects of Continuous Anterior Chest Compression
Acronym: StrapVent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP211357
Record Dates: First submitted 2022-08-08; First posted 2023-05-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Evaluable
Keywords: ARDS : Acute Respiratory Distress Syndrome; CACC : Continuous Anterior Chest Compression; VILI : Ventilator-Induced Lung Injury; ARDS,Human: Adult Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A description of each arm of the clinical trial that indicates its role in the clinical trial (Experimental): Arm 1 Description:
  The study will consitent of recording the measurments of ventilatory settings, respiratory mechanics, flow and pressure curves, gaz exchange, haemodynamics and ventilation distribution in 5 consecutive conditions in adult patients with moderate to severe ARDS :
  * After 16 hours of prone position
  * In supine position 1 hour after the prone position
  * 15mn after CACC with a pressure equal to the one observed in the prone position
  * 15mn after CACC with a pressure set at 60 - 80 cmH20
  * 15mn after taking of the CACC
  Interventions: Device: Continuous anterior chest compression

INTERVENTIONS:
Device: Continuous anterior chest compression — Patients with severe to moderate ARDS who were placed in prone position by the attending physician :
  * First CACC : the applied pressure is equal to the one observed in the prone position
  * Second CACC : The applied pressure is set at 60 - 80 cmH20

SUMMARY:
The aim is to test the physiological effects of continuous anterior chest compression in patients with severe to moderate ARDS.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is usually characterized by inhomogeneous lesions, leading to an inhomogeneous distribution of the mechanical ventilation with the following several deleterious effects: atelectrauma of dependent posterior areas and overdistension in the anterior ones. Therefore, the gold standard treatment is to prevent VILI with lung protective ventilation : low tidal volume, high positive end expiratory pressure and prone positioning which is a technique that reduces mortality. Prone positioning has several beneficial effects : it relieves cardiac compression of the supporting lung, it stiffens the anterior chest wall thus limiting the risk of overdistension of anterior areas and promotes recruitment of non-dependent posterior pulmonary units. The overall effect is a more uniform distribution of transpulmonary pressures and improved ventilation to perfusion ratios.

Similar to prone positioning, continuous anterior chest wall compression stiffens the anterior chest wall. The investigators hypothesize that such reduction in anterior chest wall compliance may protect against overdistension and promote the redistribution of the ventilation in posterior areas.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Intubated moderate and severe ARDS according to the Berlin definition (PaO2/FiO2 ratio <= 200 mmHg)
* The patent must be sedated and paralyzed
* Informed consent from patient or family members

Exclusion Criteria:

* Extracorporeal membrane oxygenation (ECMO)
* Pneumothorax
* Thoracic trauma during the last 3 months
* Refractory shock
* Contraindication to EIT monitoring (e.g. burns, pacemaker, thoracic wounds limiting electrode belt placement)
* Pregnancy
* Any contra-indication to esophageal manometry (less than one month esophagus surgery, bronchopleural or esotracheal fistula, latex allergy)
* No social care
* Adults under Guardianship, curatorship or protection of the court

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
The end inspiratory transpulmonary pressure (PL-insp) in centimetre of water | Through study completion (up to 6 hours)
  The transpulmonary pressure will be measured by using an esophageal catheter connected to a differential pressure transducer. The PL-insp will be calculated using the ratio between the elastance of the lung (El) and of the respiratory system (Ers) expressed in centimetre of water thanks to this formula PL-insp = Plateau pressure x (El/Ers). The PL-insp between the different protocol conditions will be compared (After 16 hours of prone position, in supine position, 15mn after CACC with a pressure equal to the one observed in the prone position, 15mn after CACC with a pressure set at 60 - 80 cmH20, 15mn after taking off the CACC in supine position ). CACC will be considered protective if there is a decrease in Pl-insp.

SECONDARY OUTCOMES:
Regional pulmonary compliances in centimetre of water | Through study completion (up to 6 hours)
  Evaluation and comparison of pulmonary compliances in the different regions of interest (ROI) measured by Electrical Impedance Tomography (EIT) in the different protocol conditions.
Lung mechanics : Airways pressure, Flow curves and Esophageal pressure | Through study completion (up to 6 hours)
  Airways pressure (Paw) will be measured in cmH2O and recorded by the mean of a differential pressure transducer.
  Flow curves will be measured in L/mn and recorded by the mean of a pneumotachograph connected to the ventilator circuit.
  Esophageal pressure (Pes) will be measured in cmH2O and recorded thanks to an esophageal balloon catheter introduced in the mid-esophagus of the patient and connected to differential pressure transducer.
  Evaluation and comparison of respiratory mechanics in the different protocol conditions.
Pulmonary ventilation distribution in percentage | Through study completion (up to 6 hours)
  Evaluation and comparison of the distribution of ventilation in the different regions of interest (ROI) measured by Electrical Impedance Tomography (EIT) in the different protocol conditions
Recruitment-to-inflation (R/I) ratio | Through study completion (up to 6 hours)
  Evaluation and comparaison of R/I in the different protocol conditions
Hemodynamics | Through study completion (up to 6 hours)
  Heart rate will be expressed in beats per minute, arterial blood pressure will be expressed in millimetre of mercury and norepinephrine perfusion will be expressed in milligrams per hour.
Arterial blood gazes (ABG | Through study completion (up to 6 hours)
  pH, PaCO2 and PaO2 will be measured by standard clinical technique using the ICU blood gaz analyzer. PaCO2 and PaO2 will be expressed in millimetre of mercury.
Incidence of CACC adverse events | Through study completion (up to 6 hours)
  CACC will be interrupted if :
  * Reduction in oxygen saturation (SpO2) beneath 88% despite FiO2 optimisation.
  * Reduction in mean arterial pressure beneath 60 mmHg
  * Increase in norepinephrine perfusion beyond 0.5 mg/h
End expiratory lung impedance (EELZ) expressed in arbitrary units | Through study completion (up to 6 hours) ]
  Evaluation and comparison of EELZ using EIT in the different protocol conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CARTEAUX, MD, PhD, Principal Investigator — APHP
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France